CLINICAL TRIAL: NCT05258916
Title: Feasibility and Contribution of a Nurse Consultation in the Follow-up of At-risk Newborn at Maternity Discharged: 3-year Experience in a Tertiary Center.
Brief Title: Contribution of a Nurse Consultation in the Follow-up of At-risk Newborn at Maternity Discharged
Acronym: NURCO-NEO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0001
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: At-risk Newborn
Keywords: nurse consultation; at-risk newborn; PED visits; PED hospitalizations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Nurse consultation — nurse consultation carried out within two weeks after maternity discharged

SUMMARY:
The postnatal period is a critical phase involving important physiological, psychological and social changes. Pediatric nurses could be a crucial actor in the follow-up of at-risk newborn, in collaboration with other health professionals and contribute to a reduction in pediatric emergency department (PED) visits and/or hospitalization in first weeks of life. To describe population of at-risk newborns who attended a nurse consultation after discharge from a type 3 maternity hospital and to evaluate the impact of a post-hospitalization nurse consultation for at-risk newborns on PED visits and hospitalizations.

DETAILED DESCRIPTION:
The postnatal period is a critical phase involving important physiological, psychological and social changes. In 2013, WHO recommends at least three postnatal contacts on day 3, between days 7 and 14, and six weeks after birth. Despite these recommendations, pediatric emergency department (PED) visits for newborns are constantly increasing. Some studies have shown that most of these visits were related to nonserious diseases, mainly due to a lack of knowledge and information. At the same time, some high-risk newborns have been identified as likely to be admitted to PED and subsequently hospitalized. All these findings highlight the great need for education and parental support by health staff from the time of maternity discharged, particularly when certain high-risk conditions are identified.

In France, guidelines on maternity discharge after childbirth include pediatric nurses as professionals involved in postnatal follow-up. Pediatric nurses could be a crucial actor in the follow-up of at-risk newborn, in collaboration with other health professionals and contribute to a reduction in PED visits and/or hospitalization in first weeks of life.

ELIGIBILITY:
Inclusion Criteria:

* All at-risk newborns addressed to nurse consultation after discharge from maternity hospital.
* All at-risk newborns discharged home after hospitalization at birth in the neonatal medicine department.

Exclusion Criteria:

* Newborns discharged with home hospitalization
* Consultation for hearing screening, blood testing or injection (vaccines or palivizumab).
* Newborns referred by pediatrics department, PED or by exterior professionals.
* Non-at-risk newborns hospitalized for other reasons (biological anoxia, early neonatal bacterial infection, transient tachypnea, monitoring)

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Neonates born and/or hospitalized at a tertiary center, Centre Hospitalier Sud Francilien, Corbeil Essonnes, France defined as follow.
Sampling Method: Probability Sample
Enrollment: 1330 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
PED visits at 2 weeks | 2 weeks after discharge of maternity hospital
  Number and causes of PED visits

SECONDARY OUTCOMES:
PED visits at 3 months | 3 months after discharge of maternity hospital
  Number and causes of PED visits
Hospitalization | 3 months after discharge of maternity hospital
  Number and causes of hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No